CLINICAL TRIAL: NCT02145481
Title: Decisional Quality for Patients With Stable Coronary Artery Disease
Brief Title: Decisional Quality for Patients With Coronary Artery Disease
Acronym: DeQCAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Missouri, Kansas City (Other); Mid America Heart Institute (Other); Emory University (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HL114918-01A1
Record Dates: First submitted 2014-05-15; First posted 2014-05-23 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; decision quality; decision making; survey; measure development; patient-centered care; cardiology; heart disease
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Survey development (No Intervention): Patients with coronary artery disease will be given a survey to complete assessing their knowledge, communication with physicians, involvement, and treatment preferences after completing the treatment decision-making process.
- Decision Aid (Experimental): Patients with stable coronary artery disease will be given a decision aid to review prior to making a treatment decision.
  Interventions: Behavioral: Decision Aid
- CAD Education (Active Comparator): Patient with coronary artery disease will be given a general educational handout on coronary artery disease.
  Interventions: Behavioral: CAD Education

INTERVENTIONS:
Behavioral: Decision Aid — Decision aid describing treatment choices for patients with coronary artery disease.
  Arms: Decision Aid
Behavioral: CAD Education — Education for patients with coronary artery disease
  Arms: CAD Education

SUMMARY:
The objective of the DeQCAD study is to measure the quality of the decision-making process for patients with coronary artery disease (CAD) and Acute Coronary Syndrome (ACS) who are making treatment decisions. In particular, this study is seeking to answer: a) How informed are patients about their treatment choices, b) are patients participating in the decision-making process as much as they would like to, and c) do the treatment decisions made match patients' preferences?

DETAILED DESCRIPTION:
For patients with coronary artery disease (CAD), having a stent (or percutaneous coronary intervention or PCI) involves both risk and inconvenience, and thus it represents a classic "preference-sensitive" situation, in which treatment decisions should be aligned with the patient's preferences.

In this project the investigators will develop the first comprehensive, patient-reported measure of decisional quality for CAD that is feasible to implement in a variety of settings. The investigators will accomplish this by: 1) Identifying the key elements to capture decisional quality and identifying candidate questions to address these elements, using patient and expert feedback; 2) Pilot testing a preliminary instrument in a diverse patient population to assess measurement properties and select a reduced set of candidate questions for further testing; and 3) Establish the reliability and validity of a new comprehensive decisional quality measure for single and repeated examinations. This will result in a multidimensional decisional quality instrument for patients with CAD that will be ready for implementation into routine care.

ELIGIBILITY:
Inclusion criteria:

1. Patients ≥ 18 years old
2. Able to answer survey questions in English
3. Diagnosis of coronary artery disease in one of the following categories:

   1. Stable CAD group

      * Meets any 1 of the following 3 criteria for stable CAD: 1) The patient has a clinical diagnosis or prior history of CAD; 2) Angina without change in frequency or pattern for the 6 weeks prior to enrollment; 3) Angina is controlled by rest and/or sublingual/oral/transcutaneous medications.
      * Accelerating pattern of stable angina with: 1) no ECG changes at rest; 2) no cardiac marker evidence of myocardial necrosis (e.g., elevated troponin or CK-MB); 3) scheduled for elective or urgent cardiac catheterization after being evaluated in the outpatient setting (i.e., not from the emergency department or inpatient hospitalization).
   2. Acute coronary syndrome group • Acute coronary syndrome where there is cardiac marker evidence of myocardial necrosis (e.g., elevated troponin or CK-MB) without new ST-segment elevation. Includes non-ST-elevation MI (NSTEMI).

Exclusion criteria:

1. Diagnosis of ST-elevation MI (STEMI), defined as an acute coronary syndrome in which there is cardiac marker evidence of myocardial necrosis (eg, positive troponin or CK-MB) and new (or presumably new if no prior ECG is available) ST-segment elevation or left bundle branch block on the admission ECG.
2. Unstable angina, defined as 1) Angina occurring at rest and prolonged, usually ≥ 10 minutes; 2) New onset angina of at least CCS classification III severity (i.e., marked limitation of ordinary physical activity - angina occurs on walking 1 to 2 blocks on the level and climbing 1 flight of stairs in normal conditions and at a normal pace); 3) no cardiac marker evidence of myocardial necrosis (e.g., negative troponin or CK-MB).
3. Acute coronary syndrome with hemodynamic instability (e.g., cardiogenic shock, hypotension, cardiac arrest, ongoing or recurrent chest pain, dynamic ST change).
4. Noncardiac chest pain: Pain in the chest, neck, arms, or abdomen (or other clinical manifestation) not clearly exertional or not otherwise consistent with pain or discomfort of myocardial ischemic origin.
5. Cognitive impairment such that the patient cannot give informed consent for himself or herself.
6. Unable to answer survey questions in English.
7. Unavailable for follow-up surveys

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 677 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Decision quality survey | 3 months post baseline
  Decision quality for coronary artery disease patients making treatment decisions. Our primary outcome measure is the quality of the decision making process for patients with coronary artery disease including knowledge, communication, involvement, and treatment preferences measured at Baseline and 2 weeks during the pilot test phase, and Baseline, 1 month, and 3 months during the field test phase.

CONTACTS AND LOCATIONS:
Overall Officials: R. Adams Dudley, MD, MBA, Principal Investigator — University of California, San Francisco
Locations (4):
- United States (4):
  - University of California, San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia
  - Truman Medical Center, Kansas City, Missouri
  - St. Luke's Mid-America Heart Institute, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No